CLINICAL TRIAL: NCT05958628
Title: The Efficiency of Robotic Hand Exoskeleton System in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Fatma Ozturk, researcher, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MarmaraU-FTR-FO-01
Record Dates: First submitted 2023-07-16; First posted 2023-07-24 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Stroke; Hemiplegia; Exoskeleton Device; Muscle Spasticity; Quality of life
MeSH Terms: conditions — Stroke; Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Two groups; one group will receive conventional physiotherapy and one group will be operated with robotic hand exoskeleton system in addition to conventional physiotherapy.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment will be performed by a investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Participants in this group will receive a conventional physiotherapy program 3 times a week for 5 weeks, each session lasting 1 hour.
  Interventions: Other: Conventional physiotherapy
- Intervention group (Experimental): Participants in this group will receive Robotic Hand Exoskeleton System for 10 minutes in addition to 50 minutes of conventional physiotherapy 3 times a week for 5 weeks.
  Interventions: Other: Conventional physiotherapy; Other: Robotic Hand Exoskeleton System

INTERVENTIONS:
Other: Conventional physiotherapy — The treatment program was designed in line with the patients' compliance, functional capacities and rehabilitation goals as neurodevelopmental therapy based on the ability to adapt to change, reorganization and healing in the brain by focusing on neuroplasticity from neurodevelopmental treatment approaches; Proprioceptive neuromuscular facilitation techniques to increase selective and voluntary movement; functional exercises to increase motor control skills, stretching exercises for spasticity and neuromuscular electrical stimulation.
  The control group received conventional physiotherapy exercises for 45 minutes and neuromuscular electrical stimulation for 15 minutes.
Other: Robotic Hand Exoskeleton System — In the treatment applications with the robotic hand exoskeleton system, which is designed to accelerate the healing process of patients in need of hand rehabilitation, to gain motor skills, to provide strength training and to increase participation in treatment, the patient will be asked to allow the system to move the hand at adjusted angles for 10 minutes and to accompany this movement. In the applications, while the patient is sitting comfortably and safely, the patient will be asked to place the stroke-affected hand into the system. The hand of patients who may have difficulty due to the functional status of the upper extremity and the severity of spasticity will be placed with the help of the physiotherapist. The physiotherapist will be with the patient throughout the application.
  Arms: Intervention group

SUMMARY:
The aim of our study is to investigate the effects of the robotic hand exoskeleton, on the spasticity, motor control skills, level of daily living activity, quality of life and functional independence of stroke patients.

DETAILED DESCRIPTION:
Stroke is a condition that occurs as a result of an ischemic or hemorrhagic intracranial vascular event, is the third leading cause of death in the world and can lead to disability. Depending on the localization of brain damage after stroke, it is possible to talk about different prognoses and therefore different functional losses in the lower extremities, upper extremities and hand and wrist.

Today, various neurophysiological approaches, exercise strategies, electrotherapy modalities and assistive devices are used in the rehabilitation program suitable for the patient after stroke. In addition to these, robot-assisted therapy is gaining a place as an innovative approach in stroke rehabilitation with the developments in technology. Robot-assisted therapy is thought to both facilitate and intensify treatment after stroke and increase motor development.

The normal functions of the hand, which has many abilities and a complex structure, is extremely important to lead a free and active life. When the literature is examined, the success rate in the recovery of skills and functional recovery of the hand in stroke rehabilitation is low compared to the lower extremity and shoulder joint. More interventions are needed to increase the functional recovery of the hand. Studies should be conducted on robot-assisted treatment methods that allow active and passive exercises in the hand after stroke and contribute to neuroplasticity with an intensified and standardized program.

Our aim in this study is to investigate the efficacy of the Robotic Hand Exoskeleton System developed at Marmara University in order to reduce the physiotherapy process and increase the responses of patients who have partially lost their hand functions due to stroke and need rehabilitation in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with stroke by a neurologist
* At least 3 months have passed after the stroke
* Mini Mental State Examination score of at least 24
* To be able to maintain sitting balance during working with the robot,
* Having full range of motion in the metacarpophalangeal (MCP), proximal interphalangeal (PIF) and distal interphalangeal (DIF) joints,
* Spasticity in finger flexor and extensor muscles ≤ 3 according to the Modified Ashworth Scale (MAS)
* Being between the ages of 35-85

Exclusion Criteria:

* Other neurological or orthopedic problems that may affect upper extremity function,
* Cardiovascular vulnerability (severe uncontrolled hypertension, severe coronary artery disease, unstable angina)
* Behavioral and cognitive conditions that affect treatment and make compliance difficult
* Having botulinum toxin procedure in the last 6 months
* Cardiac pacemakers
* Those with skin ulcers
* Pregnancy
* History of metastatic cancer

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Frenchay Arm Test | 5 weeks
  It is a scale that evaluates the motor control skills and functions of the upper extremities of patients in a practical way and takes less than 3 minutes to perform. The patient is asked to perform 5 tasks based on activities of daily living in a sitting position with hands on the table. The maximum score on the scale is 5, with 1 point for each successful task. (The tasks the patient is asked to do are; Fixing the ruler, Holding a cylinder, Lifting the glass, Attaching the latch to the bar, Combing hair)

SECONDARY OUTCOMES:
modified ashworth scale | 5 weeks
  The modified Ashworth scale is designed to measure the resistance encountered when moving the limb passively at full range of motion. A value of 0 indicates normal muscle tone and 4 indicates the presence of intense spasticity.
Upper Limb Motor Activity Diary-28 | 5 weeks
  The Upper Extremity Motor Activity Diary-28 is a scale consisting of 28 questions that measure the amount of use of the affected upper extremity in daily activities and the quality of the activity when used, and each question is scored between 0-5. Self-care activities, some housework and some activities that can be done in community life are questioned.
Stroke impact scale version 3.0 | 5 weeks
  It was developed in 1999 to assess the quality of life and functional independence of post-stroke patients and consists of 59 questions with 8 sub-headings: strength, memory and memory, emotion, communication, activity of daily living, mobility, hand function, social participation. All questions are used to assess the difficulties experienced by the patient in the last week. The evaluation is based on 5 points. In addition to 59 questions in 8 sub-sections, it also includes a visual analog scale (0: No improvement, 100: Complete recovery) in which the patient's perception of global recovery after stroke is evaluated with 0-100 points. The score of all subcategories is summed, and the higher the total score obtained from the scale, the better the quality of life of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Öztürk, Msc, Principal Investigator — Marmara University; Gönül Acar, assoc.prof, Study Director — Marmara University
Locations (1):
- Fatma Ozturk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No